CLINICAL TRIAL: NCT07112612
Title: Application of Personalized Minimal Residual Disease in Predicting Therapeutic Efficacy in Metastatic Hormone-sensitive Prostate Cancer
Brief Title: Minimal Residual Disease Used in Predicting Therapeutic Efficacy in Metastatic Hormone-sensitive Prostate Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Sheng Tai, Chief Physician, Anhui Medical University
Other Study IDs: PJ 2024-11-47
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: MRD; Prostate Cancer; mHSPC
Keywords: minimal residual disease; MRD; PCa
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — prostate needle biopsy tissue and bone metastasis needle biopsy tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, single-center, observational study of patients with newly diagnosed metastatic hormone-sensitive prostate cancer (mHSPC). Minimal residual disease (MRD) detection is used to investigate the actual efficacy responses of mHSPC patients with different gene mutation characteristics to treatment regimens. Factors influencing efficacy are further analyzed to provide a basis for the precise clinical diagnosis and treatment of mHSPC patients.

DETAILED DESCRIPTION:
This is a prospective, single-center, observational study designed to observe the therapeutic response of metastatic hormone-sensitive prostate cancer(mHSPC) patients with different gene mutation characteristics to treatment regimens. The study will recruit 50 mHSPC patients from the First Affiliated Hospital of Anhui Medical University and design a personalized minimal residual disease (MRD) kit based on the data of the biopsy before treatment. The blood routine, biochemical indicators, sex hormone levels, prostate multi-parameter magnetic resonance imaging (Mp-MRI), quantitative whole-body bone examination, and PSMA-PET-CT examination of the study cohort patients will be recorded. During the treatment, MRD will be tested every three months, and the MRD level, blood routine, biochemical markers, sex hormone levels, and PSA levels; patients in the study cohort will undergo prostate multiparametric magnetic resonance imaging (Mp-MRI) and quantitative whole-body skeletal examination every three months. If PSA progression occurs during follow-up, the PSA recheck frequency will be customized. This prospective, observational study will explore the response efficiency of mHSPC patients with different gene mutation types to treatment regimens through MRD detection, analyze the relevant factors affecting the efficacy, and provide a basis for the precise clinical diagnosis and treatment of mHSPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and younger than 85 years;
2. Patients diagnosed with prostate acinar adenocarcinoma, ductal adenocarcinoma, or intraductal carcinoma by pathological histology;
3. Patients with clear distant metastases found by imaging (in accordance with RECIST criteria);
4. Patients with locally advanced (N1) and metastatic (M1) prostate cancer at diagnosis.
5. Patients who have not received endocrine therapy or other systemic anti-tumor treatments in the past;
6. ECOG score of 0-2 points, with an expected survival period of more than 6 months;
7. Patients with normal organ function;
8. Routine blood test (no blood transfusion or blood products within 14 days):

   Hemoglobin (HGB) ≥ 90g/L; Absolute neutrophil count (ANC) ≥ 1.5×109/L (1500 /mm3); Platelet count (PLT) ≥ 75×109/L; White blood cell count (WBC) ≥ 3×109/L;
9. Biochemical examination:

   Total bilirubin (TBIL) ≤ upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ULN; Creatinine clearance (CCr) ≥ 30ml/min; (Cockcroft-Gault formula);
10. Coagulation function: prothrombin international normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) < 4 seconds;
11. Patients agree to sign informed consent and are able to attend scheduled study visits, provide clinical information, and cooperate with other study procedures.

Exclusion Criteria:

* (1) Patients diagnosed with neuroendocrine/small cell prostate cancer by pathological histology; (2) No clear distant metastasis was found by imaging (in accordance with RECIST criteria); (3) Patients with a history of previous treatment: including neoadjuvant and adjuvant therapy; (4) The samples submitted for examination failed to meet the quality control requirements.

  (5) Patients with combined endocrine, metabolic system diseases or other serious digestive system diseases; (6) Patients with combined chronic hepatitis, cirrhosis, chronic nephritis, renal insufficiency and other diseases; (7) Patients with a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; (8) Patients with a history of other malignant tumors; (9) Patients enrolled in other clinical trials; (10) Patients unable to obtain the clinical information required for the study (e.g., patients lost to follow-up); (11) Other situations that the researchers consider unsuitable for enrollment.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with metastatic hormone-sensitive prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
minimal residual disease(MRD) positive rate | baseline
  The probability of patients in the study cohort testing positive using the minimal residual disease (MRD) test kit.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2026-01-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT07112612/Prot_SAP_002.pdf
  • Informed Consent Form (2026-01-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT07112612/ICF_003.pdf